CLINICAL TRIAL: NCT05809661
Title: İnvestigation of the Effect on Nurse Navigation Program on Compliance, Quality of Life and Prevention of Complications in Patients With Stoma
Brief Title: Implementation of the Nurse Navigation Program
Acronym: rct
Status: Completed | Type: Observational
Sponsor: Kilis 7 Aralik University (Other)
Responsible Party: Principal Investigator, Gülistan YURDAGÜL, prelector, Kilis 7 Aralik University
Other Study IDs: 19862023
Record Dates: First submitted 2023-01-31; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Intestinal Cancer
Keywords: Nursing, Navigation Program, Stoma, Compliance
MeSH Terms: conditions — Intestinal Neoplasms; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- deney grubu: adult patients with intestinal stoma: The first interview: the patients were informed about the purpose of the study and signed informed consent form. The training booklet was delivered to them. Their contact information was obtained and the contact information of the researcher (navigator nurse) was shared with them. They were told that they could call the navigator nurse, send a message to him/her, take a photo of the stoma and share it with his/her when necessary, when they had physical, social, and psychological problems in the stoma or in line with their changing needs. In the next 3 months, they were informed about the applications to be made within the scope of the study (phone calls, information messages and videos, guidance and appointment planning). Appointment was scheduled for the next interview in 3 months.
  .
  Interventions: Behavioral: implementation of the nurse navigation program
- kontrol grubu: adult patients with intestinal stoma: The first interview: the patients were informed about the purpose of the study and signed informed consent form. All of the data collection tools were filled out. Their questions about stoma care were answered. Training booklet was handed down to them. An appointment was scheduled for the next interview 3 months later.
  The second interview (3 months after the first interview): A few days before the interview, they were called up and reminded of their appointment. The relevant forms were filled out with them at the end of the 3rd month. Their questions about stoma care were answered. An appointment was scheduled for the next interview 3 months later.

INTERVENTIONS:
Behavioral: implementation of the nurse navigation program — Adult patients with intestinal stoma were contacted continuously for 6 months.
  Groups: deney grubu

SUMMARY:
This study was conducted as a randomized controlled intervention study with repetitive measurements in a pretest-posttest order to examine the effect of nurse navigation program on compliance, quality of life and prevention of complications in patients with intestinal stoma. The study was completed with 30 experimental and 28 control group patients with intestinal stoma in six hospitals, two of which are training and research hospitals, located in Gaziantep city center, between January 1 and December 31, 2021. While counseling, remote support, written and visual trainings, informative messages, phone calls, and appointment scheduling were applied to the patients in the experimental group within the scope of the nurse navigation program, the patients in the control group received standard care

DETAILED DESCRIPTION:
This study was conducted as a randomized controlled intervention study with repetitive measurements in a pretest-posttest order to examine the effect of nurse navigation program on compliance, quality of life and prevention of complications in patients with intestinal stoma. The study was completed with 30 experimental and 28 control group patients with intestinal stoma in six hospitals, two of which are training and research hospitals, located in Gaziantep city center, between January 1 and December 31, 2021. While counseling, remote support, written and visual trainings, informative messages, phone calls, and appointment scheduling were applied to the patients in the experimental group within the scope of the nurse navigation program, the patients in the control group received standard care. The patients were evaluated using the Patient Information Form, Stoma Complications Evaluation Form, Stoma-Related Problems Experienced Form, Ostomy Compliance Scale, and Stoma Quality of Life Scale at the first interview, at the third and sixth months.

ELIGIBILITY:
Inclusion Criteria:with intestinal stoma

* Having no mental handicap or perception problems and no communication difficulties
* No psychiatric disease
* 18 years old and over
* literate
* Capable of using a smartphone
* No vision and hearing problems
* Those who have the physical ability to change the stoma bag themselves.
* Patients with intestinal stoma for a maximum of two months were included in the study.

Exclusion Criteria:

* After agreeing to participate in the research, wanting to leave,

  * Those who died during the research process,
  * The stoma was closed during the research process,
  * Patients whose communication could not be maintained during the research process

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with intestinal stoma
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
stoma compliance | 6 month
  stoma compliance scale

SECONDARY OUTCOMES:
life quality | 6 month
  quality of life scale

CONTACTS AND LOCATIONS:
Overall Officials: nuran tosun, prof, Study Director — nuran.tosun@hku.edu.tr
Locations (1):
- Kilis 7 Aralık Üniversitesi, Kilis, Turkey (Türkiye)